CLINICAL TRIAL: NCT01783210
Title: Pregnancy Complications in Women With BMI>25 kg/m2 Enrolled in a Healthy Lifestyle and Eating Habits Program: a Randomized Controlled Trial.
Brief Title: Pregnancy Complications in Women With BMI>25 kg/m2 Enrolled in a Healthy Lifestyle and Eating Habits Program
Acronym: TLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Prof. Fabio Facchinetti, Chairman of Obstetrics and Gynecology Unit, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4043/CE
Record Dates: First submitted 2013-01-28; First posted 2013-02-04 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Maternal Obesity Complicating Pregnancy, Birth,or Puerperium; Gestational Diabetes Mellitus in Pregnancy, Diet- Controlled; Exercise Addiction; High-Risk Pregnancy; Dietary Modification
MeSH Terms: interventions — Pregnancy; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TLC(Therapeutic Lifestyle Changes) group (Experimental): Intervention: "Specific Therapeutic Lifestyle Changes program in pregnancy". TLC Program includes a diet (with a specific amount of calories and macronutrients) and a mild physical activity.
  Interventions: Behavioral: Specific Therapeutic Lifestyle Changes program in pregnancy
- Control group (Other): Intervention: "Dietary and behavioral counselling in pregnancy". The Control group receives only a simple nutritional booklet about a lifestyle and healthy diet during pregnancy without explicit caloric restriction, in accordance with Italian Guidelines for a healthy diet during pregnancy, compatible with a recommended nutritional intake.
  Interventions: Behavioral: Dietary and behavioral counselling in pregnancy

INTERVENTIONS:
Behavioral: Specific Therapeutic Lifestyle Changes program in pregnancy — TLC Program includes diet and mild physical activity. The TLC comprises 1500 kcal/day (3 main meals and 3 snacks) composed of 55% carbohydrate, 20% protein, and 25% fat. The dietitian adds an 200 kcal/day for obese or 300 kcal/day for overweight. The exercise intervention is focused on increasing walking. All participants are advised to participate in 30 min of moderate intensity activity at least 3 days a week. Subjects wear a pedometer waist during walking session for the assessment of the adherence to the physical activity program. Women are told to consider using the "talk test" (being able to maintain a conversation during activity) to monitor exercise intensity, and to record the frequency and duration of the activity on a diary . Follow-up is performed at 16, 20, 28, 36 weeks.
  Arms: TLC(Therapeutic Lifestyle Changes) group
Behavioral: Dietary and behavioral counselling in pregnancy — The Control group receives only a simple nutritional booklet about a lifestyle and healthy diet during pregnancy without explicit caloric restriction, in accordance with Italian Guidelines for a healthy diet during pregnancy, compatible with a recommended nutritional intake.
  30 minutes counseling session about the appropriate gestational weight gain (GWG) at term for each different BMI category is performed. Moreover, the importance of the limited GWG for preventing unfavorable maternal-neonatal outcomes related to excessive weight gain is explained. Women are scheduled to have a follow-up at 16, 20, 28, 36 weeks.
  Arms: Control group

SUMMARY:
The investigators evaluate if changing eating habits and introducing a correct lifestyle in women with BMI >25 Kg/m2 would improve unfavorable maternal-fetal outcomes associated with excessive weight gain (EWG) during pregnancy. To pursue these goals, eligible women are randomly assigned to no intervention (Control group) that receive only a simple nutritional booklet about lifestyle and healthy diet during pregnancy without explicit caloric restriction or the Therapeutic Lifestyle Changes Program (TLC group) that receive a caloric restriction (1500 Kcal/day divided in3 main meals and 3 snacks + 300 kcal/die for overweight or 200 kcal/die for obese women submitted to energy expenditure program) associated to a mild physical activity (30 minutes at least 3 days/week) The investigators use a tool that could easily and practically evaluate not only total GWG at term, but also changes in maternal body composition: the bioimpedance analyzer.

DETAILED DESCRIPTION:
Pregnant women, recruited from antenatal clinics, with pre-pregnancy BMI ≥ 25 kg/m2, age >18 years and single pregnancy are enrolled within 12th week at the Obstetric Unit of Policlinico Hospital of Modena.

Exclusion criteria are as follows: twin pregnancies, chronic diseases (i.e., diabetes mellitus, chronic hypertension, untreated thyroid diseases), gestational diabetes mellitus (GDM) in previous pregnancies, smoking during pregnancy, dietary supplements or herbal products known to affect body weight, other medical conditions that might affect body weight, and plans to deliver outside of the Birth Center.

At the first visit, an accurate obstetric history, family history, and personal history is collected for the assessment of exclusion criteria. The blood pressure, height and weight are measured, and the BMI is calculated.

Eligible women are randomly assigned to no intervention (Control group) or the Therapeutic Lifestyle Changes Program (TLC group). Randomization is performed using sealed envelopes(using a computer-generated random allocation). Study randomization is numbered and sealed in white envelops. Randomization occurs in consecutive order at time of the first visit. Due to study design, both gynecologist and dietitian know the allocation of the patient.

Every subject receives care in another institution (Antenatal Clinics of Modena Health program). Hence, women in both groups receive the same antenatal evaluation including two ultrasound examinations and at least 4 obstetric evaluations until term. However, referral gynecologists possibly know the allocated arm of their women.

Randomized subjects receive a 75-g 2-h Oral Glucose Tolerance Test (OGTT) at 16-18 and/or 24-28 weeks. The diagnosis of GDM is made for any glucose value exceeding the normal cut-off, as reported by the HAPO study. If OGTT is pathological, women are referred to other health care specialists.

Women randomized to both group are scheduled to have a specific follow-up for adherence to the program at 16, 20, 28, 36 weeks and 3 months after delivery also evaluating the fat mass, fat-free mass and total body water through the use of the bioimpedance analyzer. At baseline and 36 weeks each subject have to complete a Food Frequency Questionnaire (FFQ) to identify any change in eating habits. The FFQ includes questions about specific food items, such as the frequency of sauce consumption, the fat content of several food items, and seasonal consumption of fruit and vegetables. While the Control group receives only a simple nutritional booklet about a lifestyle (in accordance with Italian Guidelines for a healthy diet during pregnancy), the TLC Program includes a specific caloric restriction associated to a mild physical activity program.

The TLC diet comprises 1500 kcal/day and consists of 3 main meals and 3 snacks (breakfast, snack, lunch, snack, dinner, and evening snack) that corresponds to the baseline metabolism of a pregnant woman. The dietitian adds an amount of 200 kcal/day for obese or 300 kcal/day for overweight pregnant women submitted to physical activity program.The TLC diet has a target macronutrient composition of 55% carbohydrate, 20% protein, and 25% fat with moderately low saturated fat levels. The exercise intervention is focused on increasing walking and developing a more active lifestyle (i.e., walking rather than driving for short distances). The recommended exercise prescription for pregnant women is generally consistent with recommendations for the general adult population. However, it is important to monitor and adjust exercise prescriptions according to the woman's symptoms, discomforts, and abilities during pregnancy and be aware of contraindications for exercising during pregnancy. All participants are advised to participate in 30 min of moderate intensity activity at least 3 days a week. Subjects wear a pedometer (Omron Walking Style III HJ-203-EK) on a belt at the back of their waist during walking session for the assessment of the adherence to the physical activity program.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25 kg/m2
* age >18 years
* single pregnancy
* 1st trimester

Exclusion Criteria:

* twin pregnancies
* chronic diseases (i.e., diabetes mellitus, chronic hypertension, untreated thyroid diseases)
* Gestational diabetes mellitus in previous pregnancies
* smoking during pregnancy
* dietary supplements or herbal products known to affect body weight
* other medical conditions that might affect body weight
* to plan to deliver outside of the Birth Center.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2012-07 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Gestational diabetes mellitus. | At 16-18 and/or 24-28 weeks
  Subjects of both groups receive a 75-g 2-h Oral Glucose Tolerance Test (OGTT) at 16-18 weeks and, if negative, repeated at 24-28 weeks. The diagnosis of GDM is made for any glucose value exceeding the normal cut-off, as reported by the HAPO study. If OGTT is pathological, women are referred to other health care specialists for glycemia monitoring and evalution of further therapies, in addition to the diet.

SECONDARY OUTCOMES:
Gestational wieght gain. | At baseline, 16,20,28 and 36 weeks, at delivery and 3 months after delivery.
  Excessive gestational wieght gain is a cause of unfavorable outcome of pregnancy. Weight gain is measured at each follow-up visit, at delivery and 3 months after delivery in both group, to evaluate possible effects of the intervention.
Pregnancy induced hypertension | At baseline, 16,20,28, 36 week and, at delivery.
  The blood pressure is assessed at each visit.
Preterm birth | between 24 and 36+6
  Both spontaneous and medically indicated preterm births are associated with obesity. We record cases of preterm birth, if it's spontaneous or not and the eventual indication.
Birthweight of the newborn | At delivery
  Obesity is associated with an increase of babies large for gestational age and macrosomia, while caloric restriction is not. We evaluted the centiles of growth and the rates of large for gestational age and small for gestational age.
Mode and timing of delivery | At delivery
  Obesity is associated with an higher incidence of caesarean delivery and operative vaginal delivery. Moreover, being associated with hypertensive disorders and gestational diabetes mellitus, it leads to an higher incidence of induction of labour, both in case of pregnancy preterm or at term.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Facchinetti, MD, Principal Investigator — Mother-Infant Department, University of Modena and Reggio Emilia, Italy
Locations (1):
- Mother-Infant Department, University of Modena and Reggio Emilia, Italy, Modena, Italy